CLINICAL TRIAL: NCT05944146
Title: The Consistency of Tracking Changes of Cardiac Output by Carotid Doppler Blood Flow and Thermodilution Technique in Cardiac Surgery Patients
Brief Title: Consistency of Carotid Doppler Blood Flow and Thermodilution Technique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Cracard
Record Dates: First submitted 2023-07-05; First posted 2023-07-13 (Actual); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Cardiac Surgery
Keywords: carotid doppler; hemodynamic
MeSH Terms: interventions — Dobutamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- cardiac surgery patients with thermodilution technique monitoring (Experimental)
  Interventions: Behavioral: passive leg raising; Drug: Dobutamine

INTERVENTIONS:
Behavioral: passive leg raising — transfer a patient from semi-recumbent position to supine position with a 45° leg lifting
Drug: Dobutamine — infusion dobutamine

SUMMARY:
Currently, the gold standard method to estimate CO is the thermodilution technique, pulmonary artery catheter (PAC) and PiCCO system included, however, the invasiveness and complexity of the thermodilution technique have limited their usefulness in many clinical scenarios. By measuring the carotid blood flow, continuous carotid doppler technique has been reported to noninvasively estimate cardiac output (CO) and other parameters related to cardiac contractility and fluid status in various cardiovascular disorders. However, to the best of our knowledge, few study has been reported to evaluate the consistency of this technique in cardiac surgery patients. The aim of this study is to evaluate the tracking ability of CO changes measured by continuous carotid doppler technique in cardiac surgery patients, use the thermodilution technique as the referenced.

ELIGIBILITY:
Inclusion Criteria:

* adult cardiac surgery patients
* with thermodilution technique monitoring
* mechanical ventilation

Exclusion Criteria:

* life threatening arrhythmia
* severe valve regurgitation
* left ventricular ejection fraction less than 30%
* patients with mechanical circulatory support

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
cardiac output by thermodilution method | 5 minutes after the patients was sedated
  measuring cardiac output using thermodilution method
cardiac output by continuous carotid doppler blood flow | 5minutes after the patients was sedated
  measuring cardiac output using continuous carotid doppler blood flow
cardiac output by thermodilution method | 2 minutes after passive leg raising
  measuring cardiac output using thermodilution method
cardiac output by continuous carotid doppler blood flow | 2 minutes after passive leg raising
  measuring cardiac output using continuous carotid doppler blood flow
cardiac output by thermodilution method | 15 minutes after termination of passive leg raising
  measuring cardiac output using thermodilution method
cardiac output by continuous carotid doppler blood flow | 15 minutes after termination of passive leg raising
  measuring cardiac output using continuous carotid doppler blood flow
cardiac output by thermodilution method | 30 minutes after dobutamine infusion
  measuring cardiac output using thermodilution method
cardiac output by continuous carotid doppler blood flow | 30 minutes after dobutamine infusion
  measuring cardiac output using continuous carotid doppler blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Zhe Luo, Study Chair — Fudan University
Locations (1):
- Zhongshan hospital Fudan University, Shanghai, Shanghai Municipality, China